CLINICAL TRIAL: NCT04455022
Title: The Volume of Blood Submitted for Culture in Neonates - a Multicentre Initiative to Improve the Value of the Test by Bedside Weighing of Blood Samples.
Brief Title: The Volume of Blood Submitted for Culture in Neonates - a Multicentre Quality Improvement Initiative.
Acronym: VOB4C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, PAWEL KRAJEWSKI, MD, Head of the Division of Neonatology, Medical University of Warsaw
Other Study IDs: VOB4C TRIAL'20
Record Dates: First submitted 2020-06-22; First posted 2020-07-02 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Neonatal Sepsis
Keywords: blood culture; newborn; blood volume; quality improvement; neonatal sepsis
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Any infant who will have a blood culture collected.: During the study period educational actions will be taken to raise the awareness of importance of collecting adequate volume of blood for culture (posters, leaflets and educational activities). The minimum volume will be defined as at least 1 ml. The paramount role of blood culture in process of ruling out newborn sepsis will be emphasized. The sample volume control by using bedside precision scale will be introduced.
  Interventions: Other: Bedside blood culture bottles weighing combined with educational interventions.

INTERVENTIONS:
Other: Bedside blood culture bottles weighing combined with educational interventions. — Educational actions will be taken to raise the awareness of importance of collecting adequate volume of blood for culture (posters, leaflets and educational activities). The minimum volume will be defined as at least 1 ml. The paramount role of blood culture in process of ruling out newborn sepsis will be emphasized. The sample volume control by using bedside precision scale will be introduced.

SUMMARY:
The study will examine if introducing the practice of checking the volume of blood culture samples in neonates by bedside weighing will improve the sensitivity of the test and increase confidence in negative results affecting the rate of extended antibiotic treatment in neonates with negative blood cultures.

DETAILED DESCRIPTION:
In the first part of the study (pre-intervention) the actual volumes of blood submitted for culture in neonates from participating neonatal units will be examined for the period of six months. The culture vials will be pre-weighted using precision scale before delivery to the units. After collecting the sample the vials will be weighted again at the time of admission to microbiology laboratory. At the end of the first phase, the results will be revealed to clinical teams and discussed. The sample volume control by using bedside precision scale will be introduced to the participating units along with educational actions to raise the awareness of importance of collecting adequate volume of blood for culture. The minimum volume of blood will be defined as at minimum 1 ml. The paramount role of blood culture in process of ruling out newborn sepsis will be emphasized. In the second phase of the study clinicians in participating centres will have an opportunity of measuring the volume of samples just after collecting. The volumes will also be independently controlled in the microbiology laboratory. The second phase will also last six months. Collected volumes will be compared to results from pre-intervention period. Clinical outcome measured by frequency of antibiotic treatment in newborn patients with negative blood culture will be compared before and after implemented changes. We hypothesize that introducing routine bedside control of the blood volume submitted for culture will result in increase confidence in negative blood culture results and decrease of antibiotic use in newborn population.

ELIGIBILITY:
Inclusion Criteria:

- Any infant in a neonatal ward who has a blood culture collected (either early-onset or late-onset sepsis suspected).

Exclusion Criteria:

- There is no exclusion criteria.

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants cared for in neonatal wards with suspected bacterial sepsis who have blood culture collected. All infants from birth to discharge will be considered eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-08 (Estimated)

PRIMARY OUTCOMES:
The volume of blood submitted for culture. | Through study completion, an average of 1 year.
  The volume of blood submitted for culture will be determined by weighing blood culture bottle before and after blood inoculation. The percentage of adequately filled blood culture bottles, i.e. at least 1 ml, will be compared between each study period.

SECONDARY OUTCOMES:
The use of systemic antibiotics. | Through study completion, an average of 1 year.
  The use of antibiotic therapy >72 hours despite negative blood culture results. The percentage of patients treated with antibiotics >72 hours despite negative blood cultures will be compared between each study period.
Blood culture false-positive rate (contamination rate). | Through study completion, an average of 1 year.
  The rate of blood culture contamination will be calculated by dividing the number of contaminated blood cultures by the total number of blood cultures collected during the study period.
Blood culture true-positive rate. | Through study completion, an average of 1 year.
  The rate of true positive blood cultures will be calculated by dividing the number of blood cultures that yield a pathogenic microorganism by the total number of blood cultures collected during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Krajewski, MD, PhD, Principal Investigator — Medical University of Warsaw
Locations (4):
- Poland (4):
  - Division of Neonatology and Neonatal Intensive Care, 1st Department of Obstetrics and Gynaecology, The Medical University of Warsaw, Warsaw, Warszawa
  - Department of Neonatology, Orlowski Public Teaching Hospital, Centre of Medical Postgraduate Education, Warsaw
  - Neonatal Unit, Holy Family Hospital, Warsaw
  - Specialistic Hospital 'Inflancka', Warsaw

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be available, after deidentiﬁcation. The study protocol will also be available. These documents will be accessible to anyone who provides a methodologically sound proposal immediately following publication with no end date.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who provides a methodologically sound proposal.

REFERENCES:
- [Background] Puopolo KM, Benitz WE, Zaoutis TE; COMMITTEE ON FETUS AND NEWBORN; COMMITTEE ON INFECTIOUS DISEASES. Management of Neonates Born at >/=35 0/7 Weeks' Gestation With Suspected or Proven Early-Onset Bacterial Sepsis. Pediatrics. 2018 Dec;142(6):e20182894. doi: 10.1542/peds.2018-2894. PMID 30455342
- [Background] Cantey JB, Baird SD. Ending the Culture of Culture-Negative Sepsis in the Neonatal ICU. Pediatrics. 2017 Oct;140(4):e20170044. doi: 10.1542/peds.2017-0044. Epub 2017 Sep 19. No abstract available. PMID 28928289
- [Background] Mukhopadhyay S, Taylor JA, Von Kohorn I, Flaherman V, Burgos AE, Phillipi CA, Dhepyasuwan N, King E, Dhudasia M, Puopolo KM. Variation in Sepsis Evaluation Across a National Network of Nurseries. Pediatrics. 2017 Mar;139(3):e20162845. doi: 10.1542/peds.2016-2845. Epub 2017 Feb 8. PMID 28179485
- [Background] Stoll BJ, Hansen N, Fanaroff AA, Wright LL, Carlo WA, Ehrenkranz RA, Lemons JA, Donovan EF, Stark AR, Tyson JE, Oh W, Bauer CR, Korones SB, Shankaran S, Laptook AR, Stevenson DK, Papile LA, Poole WK. Late-onset sepsis in very low birth weight neonates: the experience of the NICHD Neonatal Research Network. Pediatrics. 2002 Aug;110(2 Pt 1):285-91. doi: 10.1542/peds.110.2.285. PMID 12165580
- [Background] Garber SJ, Puopolo KM. Prevention of Central Line-Associated Bloodstream Infections Among Infants in the Neonatal Intensive Care Unit. 2015;16(4):e211-e20.
- [Background] Shoji K, Tsuboi N, Arakawa R, Ide K, Mikami M, Kato A, Miyairi I. Continuous Monitoring and Feedback Optimizes Blood Volume Inoculated Into Culture Bottles in the Pediatric Intensive Care Unit. J Pediatric Infect Dis Soc. 2019 May 11;8(2):166-169. doi: 10.1093/jpids/piy061. PMID 30010914
- [Background] Schelonka RL, Chai MK, Yoder BA, Hensley D, Brockett RM, Ascher DP. Volume of blood required to detect common neonatal pathogens. J Pediatr. 1996 Aug;129(2):275-8. doi: 10.1016/s0022-3476(96)70254-8. PMID 8765627
- [Background] Connell TG, Rele M, Cowley D, Buttery JP, Curtis N. How reliable is a negative blood culture result? Volume of blood submitted for culture in routine practice in a children's hospital. Pediatrics. 2007 May;119(5):891-6. doi: 10.1542/peds.2006-0440. PMID 17473088
- [Background] Buttery JP. Blood cultures in newborns and children: optimising an everyday test. Arch Dis Child Fetal Neonatal Ed. 2002 Jul;87(1):F25-8. doi: 10.1136/fn.87.1.f25. PMID 12091285
- [Background] Khare R, Kothari T, Castagnaro J, Hemmings B, Tso M, Juretschko S. Active Monitoring and Feedback to Improve Blood Culture Fill Volumes and Positivity Across a Large Integrated Health System. Clin Infect Dis. 2020 Jan 2;70(2):262-268. doi: 10.1093/cid/ciz198. PMID 30873522
- [Background] Cattoir L, Claessens J, Cartuyvels R, Van den Abeele AM. How to achieve accurate blood culture volumes: the BD BACTEC FX blood volume monitoring system as a measuring instrument and educational tool. Eur J Clin Microbiol Infect Dis. 2018 Sep;37(9):1621-1626. doi: 10.1007/s10096-018-3291-x. Epub 2018 Jun 7. PMID 29882176
- [Background] Shim H, Kim K, Uh Y, Seo D, Kim H, Yoon Y. The Development and Evaluation of Blood Volume Measuring System for Blood Culture Quality Improvement. Journal of Testing and Evaluation. 2012;40.
- [Background] Libertin CR, Sacco KA, Peterson JH. Education and coaching to optimise blood culture volumes: continuous quality improvement in microbiology. BMJ Open Qual. 2018 Jul 21;7(3):e000228. doi: 10.1136/bmjoq-2017-000228. eCollection 2018. PMID 30057953
- [Background] Birkhamshaw E, Winzor G. Increasing the volume of blood received in adult paired blood culture bottles at a regional public health laboratory: results of a quality improvement project to optimise the diagnosis of bacteraemia. Infect Prev Pract. 2019 Apr 19;1(1):100007. doi: 10.1016/j.infpip.2019.100007. eCollection 2019 Mar. PMID 34368673
- [Background] Ohnishi T, Kamimaki I, Kobayashi R, Nakatogawa K, Amemiya A, Mishima Y, Asato S, Shikoro N, Nakazawa M. Verification of blood volume for blood culture and detection rate in pediatrics. J Infect Chemother. 2020 May;26(5):471-474. doi: 10.1016/j.jiac.2019.12.008. Epub 2019 Dec 31. PMID 31899078
- [Background] Singh MP, Balegar V KK, Angiti RR. The practice of blood volume submitted for culture in a neonatal intensive care unit. Arch Dis Child Fetal Neonatal Ed. 2020 Nov;105(6):600-604. doi: 10.1136/archdischild-2019-318080. Epub 2020 Mar 20. PMID 32198199